CLINICAL TRIAL: NCT01464645
Title: Prospective Multicenter Open Label Study Examining the Short-term Safety and Efficacy of the Modular Revision Hip System (MRHS)
Brief Title: Post-Market Study of the Modular Revision Hip System
Acronym: MRHS
Status: Terminated | Type: Observational
Sponsor: Encore Medical, L.P. (Industry)
Collaborators: DJO Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: PS-804
Record Dates: First submitted 2011-11-02; First posted 2011-11-03 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2017-02

CONDITIONS: Aseptic Loosening; Osteolysis; Traumatic Fracture; Failed Total Hip Implant
MeSH Terms: conditions — Osteolysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Primary: Post Market Study
  Interventions: Device: Modular Revision Hip System

INTERVENTIONS:
Device: Modular Revision Hip System — Hip System that is indicated for patients whose bone stock is of poor quality or inadequate for other reconstruction techniques as indicated by deficiencies of the femoral head, neck or portions of the proximal femur.
  Other Names: MRHS

SUMMARY:
The purpose of this study is to examine the short term efficacy of the MRH system as well as determine if operating room time is decreased using this simple, two-tray system.

DETAILED DESCRIPTION:
The main goal of Revision Total Hip Arthroplasty (THA) is to restore the patient's hip function by repairing the patient's kinematics. However, a revision hip surgery represents a challenge for even the most experienced surgeon. Loss of bone stock, joint stability, infection, fracture, trochanteric non-union, and difficulty in implant or cement removal are all potential issues that a surgeon must consider for each presenting patient. These challenges require hip implant systems to provide an intraoperative flexibility that is not normally required for primary THA. The Lima Modular Revision Hip System uses modular stem and neck components to allow for surgical versatility when selecting leg length, offset and version. The purpose of this study is to examine the short term safety and efficacy of the Modular Revision Hip System (MHRS) using radiologic success and Harris Hip Scores as endpoints. The study will take place at multiple sites across the United States and will include only subjects who meet the indications for use criteria for the Modular Revision Hip system and who are candidates for revision hip replacement surgery. Target enrollment will be 200 subjects with up to 25 subjects at 15 sites across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for revision hip arthroplasty
* Subject must have either poor bone stock or deficiencies of the femoral head, neck or portions of the proximal femur
* Subject's hip joint must be anatomically and functionally suited to receive the hip implant
* Subject must have a body mass index of 40.00 or less (BMI) ≤ 40.00 at time of consent
* Subject must be willing and able to sign the informed consent and follow study procedures
* Subject must be 18 years of age or older (≥ 18) at the time of consent
* Subject must be willing to return for all study visits
* Subject (female) must not be pregnant at time of surgery

Exclusion Criteria:

* Subject must not be receiving a primary hip replacement
* Subject has a mental condition(s) that may interfere with the subject's ability to give an informed consent or willingness to fulfill the study requirements (i.e., severe mental retardation such that the Subject cannot understand the informed consent process, global dementia, prior strokes that interfere with the Subject's cognitive abilities, senile dementia, and Alzheimer's Disease)
* Subject has a condition that places excessive demand on the implant including high levels of physical activity (i.e. competitive sports, heavy physical labor)
* Subject has a BMI >40.00
* Subject is skeletally immature
* Subject has osteomyelitis
* Subject has loss of ligamentous structures
* Subject is a prisoner
* Subject is pregnant
* Subject has an active infection or sepsis at time of surgery
* Subject has a history of alcoholism or other addictions (current)
* Subject has muscular, neurological or vascular deficiencies which compromise the affected extremity (i.e., Parkinson's Disease, Syringomyelia and Multiple Sclerosis, Charcot joints)
* Subject has known materials sensitivity (to metals)
* Subject has a physical condition that would eliminate or tend to eliminate adequate implant support or prevent the use of an appropriately-sized implant
* Subject is unwilling to modify post-operative physical activities
* Subject is younger than 18 years of age (<18) at the time of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects will be at least 18 years of age at the time of consent and meet the inclusion criteria for a total hip revision arthroplasty due to poor bone stock, or due to deficiencies of the femoral head, neck or portions of the proximal femur.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Harris Hip Score Evaluation | 2 year
  The Harris Hip Score was developed to evaluate hip function in patients with traumatic disorders of the hip, but it is now commonly used to follow patients after surgery for a degenerative disorder of the hip (Harris et al., 1969). The score is broken down into 4 areas (pain, function, deformity and range of motion), with the best possible score being 100. 44 points are allotted for pain, 47 for mobility/function, 5 for range of motion and 4 for absence of deformity. Grading for the Harris Hip Score: Excellent (90-100), Good (80-90), Fair (70-79) and Poor (<70).
Number of Participants With Radiologic Failure of Device | 2 year
  Radiographic failure is defined as a complete radiolucent line > 2mm wide at the Prosthesis/Bone Interface or a >3 Degree Migration varus/valgus or >3 mm Subsidence of the component.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Levine, M.D., Principal Investigator — Orthopedic Associates of Pittsburgh, Inc.
Locations (6):
- United States (6):
  - Orthopaedic Surgery Specialists, Burbank, California
  - Stanford Medical Center Outpatient Clinic, Redwood City, California
  - Syracuse Orthopaedic Specialists, Syracuse, New York
  - McBride Clinic, Oklahoma City, Oklahoma
  - Orthopedic Associates of Pittsburgh, Inc., Monroeville, Pennsylvania
  - Texas Institute for Hip and Knee Surgery, Austin, Texas